CLINICAL TRIAL: NCT00131690
Title: The Importance of Caffeine in Fetal Growth
Brief Title: Effect of Caffeine on Fetal Growth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Danish Epdiemiology Science Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1994/2974
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2005-10-10 (Estimated); Status verified 2005-08

CONDITIONS: Birth Weight
Keywords: Caffeine; Coffee; Randomized; Birth weight
MeSH Terms: conditions — Birth Weight

INTERVENTIONS:
Drug: Nescafé Gold Blend (exposed)
Drug: Nescafé Decaffeinated (controls)

SUMMARY:
The purpose of this study is to determine whether caffeine has any effect on birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Consumption of at least 3 cups of coffee/day at recruitment

Exclusion Criteria:

* Gestational age more than 20 weeks at recruitment
* Chronic kidney disease
* Epilepsy
* Insulin dependent diabetes
* Metabolic disorder
* Previous low birth weight delivery
* Previous preterm delivery

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200
Dates: Start 1996-04; Study Completion 2002-08

PRIMARY OUTCOMES:
birth weight
gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Olsen, Professor, Study Chair — Danish Epidemiology Science Centre
Locations (1):
- Danish Epidemiology Science Centre, Vennelyst Boulevard 6, Aarhus, Denmark

REFERENCES:
- [Derived] Bech BH, Obel C, Henriksen TB, Olsen J. Effect of reducing caffeine intake on birth weight and length of gestation: randomised controlled trial. BMJ. 2007 Feb 24;334(7590):409. doi: 10.1136/bmj.39062.520648.BE. Epub 2007 Jan 26. PMID 17259189